CLINICAL TRIAL: NCT02133768
Title: Routine Bladder Catheterisation Through Fast-track Hip and Knee Replacement - What Are the Consequences?
Status: Completed | Type: Observational
Sponsor: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Morten Homilius, MD, Lundbeck Foundation
Other Study IDs: Bladder cathererisation; Lundbeck Foundation (Other: Lundbeck Foundation)
Record Dates: First submitted 2014-04-08; First posted 2014-05-08 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe the need for re-catheterization and incidence of urological complications of routine use of perioperative fixed urinary catheter (KAD) for up to 24 hours of fast-track THA and TKA

DETAILED DESCRIPTION:
Postoperative urinary retention (POUR) is a well known complication of fast-track total hip (THA) and knee arthroplasty (TKA), and even though medical options have been attempted, bladder catheterisation remains the only well-documented capacity to prevent and / or treat POUR.

It was previously standard to use fixed urinary catheter (KAD), the first 24-48 hours postoperatively to prevent POUR by THA and TKA, while more recent studies now recommend intermittent urinary catheterization in the postoperative period.

However, there are no detailed studies with adequate follow-up, describing the consequences of using either one or the other treatment regimen of POUR by fast-track THA and TKA.

Purpose:

To describe the need for re-catheterization and incidence of urological complications of routine use of perioperative fixed urinary catheter (KAD,catheter a demure) for up to 24 hours of fast-track THA and TKA

End Points:

1. The number of patients in need of re-catheterization due POUR
2. The number of patients in which the removal of KAD was not carried out within 24 hours.
3. The number of urinary tract infections from surgery to postoperative day (POD) 30
4. The number of patients with new-onset urinary discomfort at POD 30 (Increase in IPSS score).
5. The number of urological-related readmissions (including urosepsis) within POD 30

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following criteria to be eligible to enroll in the study:

  * Age >50 years.
  * Patients scheduled for primary THA or TKA.
  * Patients who have given verbal consent to participate in the study.

Exclusion Criteria:

* Patients who meet one or more of the following criteria may not be included in the study:

  * Patients who can not cooperate with the study.
  * Patients who do not understand or speak Danish.
  * Patients who are permanent catheter carriers or use disposable bladder catheterisation.
  * Patients on hemodialysis.
  * Urine Derivative patients.
  * Pregnancy or childbirth within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participating patients may help to clarify the consequences of using fixed bladder catheterisation of patients undergoing planned deployment of an artificial hip or knee. This will provide a basis to compare the effects of these practices with other treatment regimens, such as. intermittent once-bladder catheterisation in the postoperative period, which may contribute to the prevention and treatment of POUR can be optimized for all patients.
  The study is conducted as a non-interventional, observational study and all participants will receive the department's standard treatment.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of patients needing re-catheterization | From removal of urinary catheter at first postoperative day and untill discharge from hospital
  The need for re-catheterization will be asses on a daily basis until discharge from hospital (median 3 days from surgery)

SECONDARY OUTCOMES:
Number of patients who did not get their urinary catheter removed on the first postoperative day | within the first 24 hours after surgery
Number of urinary tract infections | within the first 30 days after surgery
  Assessed on a daily basis during admision and detailed telephone interview on day 30 after surgery
Number of patients developing postoperative micturition difficulties | From day 1 to day 30 after surgery
  All patients completes a questionary preoperatively (the international prostate symptom score) and the same questionary again on day 30 after surgery.
Number of re-admission due to urological problems, including urosepsis | within the first 30 days after surgery
  assessed by telephone interview on day 30 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Morten Homilius, Principal Investigator — Department of orthopedic, Regional Hospital Holstebro
Locations (1):
- Department of Orthopedic, Holstebro, Central Jutland, Denmark

REFERENCES:
- [Derived] Bjerregaard LS, Homilius M, Bagi P, Hansen TB, Kehlet H. Indwelling urinary catheterisation may increase risk of complications in hip and knee arthroplasty. Dan Med J. 2019 Apr;66(4):A5538. PMID 30910003